CLINICAL TRIAL: NCT07252089
Title: Impact of Decision Support Tools on Amputation Decisions in Diabetic Foot Patients: A Quasi-Experimental Study
Brief Title: Development and Application of a Decision-Making Aid Tool for Amputation Surgery in Diabetic Foot Patients Based on the Ottawa Decision Support Framework
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Shiwen Hong (Other)
Collaborators: Sir Run Run Shaw Hospital (Other)
Responsible Party: Sponsor-Investigator, Shiwen Hong, ShiWen Hongª (MS)nursing department, sir run run shaw hospital,zhejiang university school of medicine.Hangzhou, Zhejiang Province, China, Zhejiang University
Organization: Zhejiang University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: SRRSH No. 0805 (2025)
Record Dates: First submitted 2025-11-19; First posted 2025-11-26 (Actual); Last update posted 2025-11-26 (Actual); Status verified 2025-11

CONDITIONS: Diabetic Foot Disease
Keywords: Diabetic Foot Amputation Decision-Making Aid Tool
MeSH Terms: interventions — Nursing Care

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Experimental group (Active Comparator): In addition to receiving routine clinical consultations and nursing care identical to the control group, the intervention group will utilize an electronic decision-making aid for diabetic foot amputation. We will design this electronic tool and deliver it to participants via a WeChat Mini Program. Patients will be instructed to spend no more than 60 minutes using the tool, with researchers supervising their sessions and providing assistance as needed. During the study period, the electronic decision-making aid will remain confidential and accessible only to the intervention group, with restricted access for physicians and non-intervention patients.
  Interventions: Procedure: Applications of Decision-Support Tools in Amputation Decision-Making for Diabetic Foot Patients
- Control group (Placebo Comparator): Patients received routine clinical consultation and nursing care before and after random assignment.
  Interventions: Procedure: Routine Clinical Consultation and Nursing Care

INTERVENTIONS:
Procedure: Applications of Decision-Support Tools in Amputation Decision-Making for Diabetic Foot Patients — In addition to receiving routine clinical consultations and nursing care identical to the control group, the intervention group will utilize an electronic decision-making aid for diabetic foot amputation. We will design this electronic tool and deliver it to participants via a WeChat Mini Program. Patients will be instructed to spend no more than 60 minutes using the tool, with researchers supervising their sessions and providing assistance as needed. During the study period, the electronic decision-making aid will remain confidential and accessible only to the intervention group, with restricted access for physicians and non-intervention patients.
  Arms: Experimental group
Procedure: Routine Clinical Consultation and Nursing Care — Patients received routine clinical consultation and nursing care before and after random assignment.
  Arms: Control group

SUMMARY:
To verify whether amputation decision-making aids can alleviate the decisional dilemma in diabetic foot patients.

DETAILED DESCRIPTION:
Through a clinical controlled study, the nurse-assisted intervention group utilized the Decision-Making Aid Tool for Amputation in Diabetic Foot Patientsto assess patients' treatment choice stages, provide disease-related knowledge, and clarify the advantages and disadvantages of different treatment options. This tool also helped patients articulate their values and preference biases. Subsequently, a questionnaire survey was conducted to evaluate decisional conflict, decisional expectations, and decisional satisfaction between the two groups, aiming to assess the tool's application efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Diabetic foot ulcers with Wagner grade 4 or higher gangrene. Diabetic foot ulcers with Wagner grade 3 accompanied by severe infection or systemic symptoms; severe local infections, or chronic osteomyelitis causing functional impairment of the limb.

Patients with lower extremity vascular disease showing progression despite systemic treatment.

IWGDF stage 3 severe infections (characterized by loss of protective sensation or peripheral arterial disease, with at least one of the following: history of foot ulcer, lower limb amputation, or end-stage renal disease).

Exclusion Criteria:

* History of psychiatric disorders with inability to cooperate during communication.

Concomitant severe complications.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 80 (Estimated)
Dates: Start 2026-05-01 (Estimated); Primary Completion 2026-10-01 (Estimated); Study Completion 2026-10-31 (Estimated)

PRIMARY OUTCOMES:
Decisional Conflict Scale，DCS | When the patient was admitted to the hospital；Three days post-surgery；One month postoperatively
  The scale consists of 16 items and has undergone standardized conversion, with a total score of 100 points. A lower score indicates a lower level of decisional conflict in patients. A score >25 suggests the presence of decisional conflict during the decision-making process, while a score >37.5 indicates potential delays in decision-making

SECONDARY OUTCOMES:
The Control Preference Scale，CPS | When the patient was admitted to the hospital；Three days post-surgery；One month postoperatively
  The scale consists of five options, categorized into three decision-making types: Proactive, Cooperative, and Passive. Decision-makers select the option that best aligns with their expectations based on their self-assessment.
The Satisfaction with Decision Scale，SWD | Three days post-surgery ；One month postoperatively
  The scale consists of 6 items, allowing decision-makers to select the hospital description that best aligns with their individual circumstances.
Decision Regret Scale,DRS | Three days post-surgery；One month postoperatively
  The scale consists of 5 items rated using a Likert 5-point rating scale, with responses ranging from "Strongly Agree" to "Strongly Disagree" assigned scores of 1 to 5 respectively. Items 2 and 4 are reverse-coded. The total score is calculated by converting the mean score of all items using the formula:
  Total Score = (Mean Score - 1) × 5 This results in a total score range of 0-20 points, where higher scores indicate greater decision regret

IPD SHARING:
Plan to Share IPD: No